CLINICAL TRIAL: NCT04308889
Title: Pro-Resolving Mediators in Acute Inflammation in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Bruce D. Levy, Professor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P000836; 2P01GM095467-06 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Inflammation; Skin; Resolution; Blister
Keywords: Specialized pro-resolving mediators
MeSH Terms: conditions — Dermatitis; Blister | interventions — Omacor; Phlebotomy

STUDY DESIGN:
Intervention Model Description: Subjects will participate in a total of 6 study visits clustered into two groups of 3 visits (baseline, 24h and 72h after blister induction) for a total of 72 hours duration. The crossover for each group of 3 visits will be separated by at least 1 week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Without Supplementation (Active Comparator): No planned dietary supplementation
  Interventions: Other: Cantharone; Other: Phlebotomy
- With Supplementation (Experimental): The subject will take 4 capsules (1gram each) of Lovaza daily at 8pm, starting the evening before blister induction and continuing until the second blister fluid has been removed.
  Interventions: Drug: Lovaza; Other: Cantharone; Other: Phlebotomy

INTERVENTIONS:
Drug: Lovaza — Lovaza contains ethyl esters of omega-3 fatty acids (EPA and DHA) obtained from the oil of several fish sources.
  Other Names: omega-3 fatty acid ethyl esters
  Arms: With Supplementation
Other: Cantharone — Cantharone is a clinical blistering agent for topical use to remove warts and molluscum contagiosum. We plan to use the drug to elicit a small skin blister and inflammatory response. This is a well described clinical inflammation research experimental model with multiple publications of its safety and utility in tracking the host inflammatory response.
Other: Phlebotomy — Subjects will have blood drawn from the antecubital vein for not more than 15mL at each visit.

SUMMARY:
The investigators are undertaking a clinical blister model with or without dietary supplementation with omega-3 fatty acids (i.e., Lovaza) to determine the role of specialized pro-resolving mediators - endogenous lipids converted from omega-3 fatty acid precursors including those in Lovaza - on inflammation parameters and their resolution.

DETAILED DESCRIPTION:
The specific aims of this study are based on the hypothesis that in health, natural pro-resolving mechanisms, including specialized pro-resolving mediators and cellular effectors, are generated to promote the resolution of acute inflammation. The specific aims are:

Aim 1. Map the formation of specialized pro-resolving mediators and their relationship to acute tissue inflammation Aim 2. Determine the influence of omega-3 fatty acids on the formation and action of pro-resolving mediators during acute inflammation.

Medical history and clinical information will be obtained from the participant's health record for study purposes to be sure that participants meet the appropriate inclusion and exclusion criteria. The phlebotomy and topical application of the cantharidin, the imaging and clinical assessment and sampling of blister exudates will be performed by Dr. Katherine Walker or Dr. Joseph Merola and clinical study team at Brigham and Women's Hospital in the Building For Transformative Medicine (3rd floor, 60 Fenwood Road, Boston, MA). The biochemical, immunological and histological analyses will be performed in the laboratories of Drs. Bruce Levy and Charles Serhan at BWH in the Building For Transformative Medicine (3rd floor, 60 Fenwood Road).

The intervention protocol will involve simultaneous topical application of 12.5 mcl 0.1% cantharidin to two sites on the volar surface of one forearm. This dose is known to elicit a consistent, safe, localized reaction entailing redness (erythema), mild tenderness and warmth at the site, 2-3 cm in diameter. Subsequently, blister exudative fluid will be removed from each blister site, one during onset phase of inflammation (24 hrs after cantharidin) and the second during resolution phase (72 hrs after cantharidin). The blister exudates will be sampled by piercing the roof of the blister with a sterile needle to collect the exudate at designated time points. The site is disinfected prior to collection of the blister exudate and subsequently protected by a wound dressing after the sample collection step.

The intervention protocol will be performed twice for each participant, under 2 distinct conditions:

1. without omega-3 fatty acid supplementation
2. with omega-3 fatty acid supplementation: the participant will take 4 capsules (1gram each) of Lovaza daily at 8pm, starting the evening before blister induction and continuing until the second blister fluid has been removed.

This study is a crossover design to evaluate the production of pro-resolving mediators and resolution of experimental inflammation with and without additional omega-3 fatty acid supplementation, and to allow each subject to serve as an internal control by undergoing blister formation in both conditions. In order to reduce the influence of repeated cantharidin blister exposures on the outcome measurements, subjects will be randomized to start with either the Lovaza arm or the non-supplementation arm of the blister protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Ages 18-64

Exclusion Criteria:

* Known acute or chronic infection
* Known acute or chronic disease of any kind
* Known allergy to fish or shellfish
* Use of any prescription medication
* Use of over-the-counter medication except multivitamins
* Use of dietary or herbal supplement except protein supplements
* Women that are pregnant, trying to become pregnant, or breastfeeding
* Any skin disease
* Known immunocompromise, HIV, or Diabetes mellitus
* History of cardiopulmonary disease
* History of upper extremity cellulitis
* Significant allergy of any kind
* Known bleeding diathesis
* History of keloid scar formation
* Forearm tattoo
* Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) during study or within 2 weeks prior to enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Specialized Pro-Resolving Mediators in Acute Inflammation | 24 hours after blister induction
  Specialized Pro-Resolving Mediators (SPMs) in a participant's peripheral blood and blister fluid will be extracted and analyzed by targeted metabolo-lipidomics with liquid chromatography - tandem mass spectrometry to identify and quantify SPMs and related bioactive lipid mediators, namely leukotrienes and prostaglandins. Note that these fatty acids and bioactive mediators in blister exudates and peripheral blood will have the same units of measure.

SECONDARY OUTCOMES:
Inflammatory Cells in Acute Blister Exudates | Change from 24 to 72 hours after blister induction
  Blister exudate fluid will be collected for determination of the presence of inflammatory cells by total cell count, and wright-giemsa staining of cytospins. Flow cytometry will be performed to confirm cell identity.
Inflammatory Cell Changes During Resolution of Acute Inflammation | Change from 24 to 72 hours after blister induction
  Blister exudate fluid will be collected for determination of cell activation by flow cytometry, including SPM receptor expression and indicators of cell death.
Peripheral Blood Inflammatory Cells During Acute Inflammation and Resolution | Change from baseline to 24 hours and then to 72 hours after blister induction
  Peripheral blood mononuclear cells will be analyzed by flow cytometry to determine activation markers, including SPM receptor expression.
Specialized Pro-Resolving Mediator Levels During Resolution of Acute Inflammation | Change from 24 hours to 72 hours after blister induction
  Specialized Pro-Resolving Mediators (SPMs) in a participant's peripheral blood and blister fluid will be extracted and analyzed by targeted metabolo-lipidomics with liquid chromatography - tandem mass spectrometry to identify and quantify SPMs and related bioactive lipid mediators, namely leukotrienes and prostaglandins. Note that these fatty acids and bioactive mediators in blister exudates and peripheral blood will have the same units of measure.

OTHER OUTCOMES:
Laser Speckled Contrast Imaging During Acute Inflammation and Resolution | Change from baseline to 24 hours and then to 72 hours after blister induction
  Local perfusion changes within the blister and surrounding/underlying skin will be determined by laser speckle contrast imaging. This qualitative assessment allows for comparisons of cellular movement in the induction and resolution phases of the blister inflammatory responses.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Levy, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The dissemination plan for the results of this study will include publication in peer-reviewed journals and presentation at scientific meetings. No IPD is planned for sharing with other researchers.